CLINICAL TRIAL: NCT04498572
Title: The Effect of Dry Needling in the Gluteus Medius Muscle With Active Physiotherapy Versus Placebo Dry Needling With Active Physiotherapy in Patients With Chronic Low Back Pain
Brief Title: The Effect of Dry Needling of the Gluteus Medius Muscle in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2393
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2021-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: two groups. research group will receive dry needling and control group will receive sham dry needling.
Who Masked: Participant
Masking Description: participants will not be aware of the group they were assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- research group (Experimental): active exercises and dry needling for the Gluteus medius muscle
  Interventions: Other: dry needling
- control group (Sham Comparator): active exercises and sham dry needling for the Gluteus medius muscle
  Interventions: Other: sham dry needling

INTERVENTIONS:
Other: dry needling — dry needling for Gluteus Medius muscle in combination with exercises
  Arms: research group
Other: sham dry needling — sham dry needling for Gluteus Medius muscle in combination with exercises
  Arms: control group

SUMMARY:
The effectiveness of dry needling of the Gluteus Medius muscle in combination with active exercises will be examined compared with sham needling with active exercises in low back pain (LBP) patients.

DETAILED DESCRIPTION:
Objectives: To examine if dry needling in combination with active physiotherapy is more effective in reducing pain and increase activity of daily living, range of motion and muscle strength in patients with chronic low back pain compared to sham dry needling in combination with active physiotherapy.

Methods: the study will include individuals with non-specific LBP over 3 months.

Subjects will be divided randomly into two research groups, both will receive physiotherapy including mobility, strengthening and stretching exercises. Intervention group, additionally to exercises, will receive dry needling to the Gluteus Medius muscle by inserting a needle to a trigger point until a visible involuntary twitch in the muscle appears. Sham needling will be applied by needling with pre-cut and smoothed needles that will not penetrate the skin.

Both groups will receive two treatments per week and up to six treatments overall, evaluation will be performed before and after the series of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Main complaint of nonspecific LBP over a 3 month period
* VAS > 3 at baseline

Exclusion Criteria:

* two or more of the following signs are present on physical examination: lower extremity weakness in a myotome distribution, decreased sensation in a dermatomal distribution, altered lower extremity deep tendon reflexes, pathological reflexes, a positive straight leg raise (SLR) test, crossed SLR or femoral nerve stretch test.
* Symptoms began immediately after a significant trauma (motor vehicle accident, fall from a height) and subjects were not been screened for possible fractures.
* Physical therapy or chiropractic treatment for LBP was provided during the 6 months prior to participation in the study or are currently being treated.
* presence of contraindication for dry needling
* pregnancy
* past back or pelvic surgery

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
change in visual analog scale (VAS) | baseline and at 3 weeks
  assessing pain on a scale from 0 (no pain) to 10 (most sever pain). Higher scores means worse outcome.
Change in Modified Oswestry Disability Index | baseline and at 3 weeks
  questionnaire to assess the disability level associated with LBP and includes 10 questions regarding activities likely to be affected by LBP. Higher scores means worse outcome.
Global rating of change | 3 weeks
  a 15-point Likert scale ranging to assess treatment success. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change in hip abductors muscle strength | baseline and 3 weeks
  muscle strength in Newton, assessed by an hand held dynamometer
Change in lumbar flexion range of motion | baseline and 3 weeks
  lumbar flexion assessment by bending forward and measuring distance of fingers from the floor

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PhD, Principal Investigator — Gali Dar, Department of Physical Therapy, University of Haifa
Locations (1):
- Haifa University, Department of PHysical Therapy, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
following study completion, a paper will be submitted to international professional journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months following end of study

REFERENCES:
- [Result] Cooper NA, Scavo KM, Strickland KJ, Tipayamongkol N, Nicholson JD, Bewyer DC, Sluka KA. Prevalence of gluteus medius weakness in people with chronic low back pain compared to healthy controls. Eur Spine J. 2016 Apr;25(4):1258-65. doi: 10.1007/s00586-015-4027-6. Epub 2015 May 26. PMID 26006705
- [Result] Dar G, Hicks GE. The immediate effect of dry needling on multifidus muscles' function in healthy individuals. J Back Musculoskelet Rehabil. 2016 Apr 27;29(2):273-278. doi: 10.3233/BMR-150624. PMID 26406203
- [Derived] Dar G, Goldberg A. Dry needling of the gluteus-medius muscle, combined with standard care, for chronic low back pain - a pilot randomized sham-controlled trial. J Man Manip Ther. 2025 Oct;33(5):392-400. doi: 10.1080/10669817.2025.2465726. Epub 2025 Feb 15. PMID 39954045